CLINICAL TRIAL: NCT07308639
Title: DATA-INSIGHT: Data Analysis for Treatment Assessment and Evaluation of New Sources for Evidence Generation in German Healthcare System
Brief Title: DATA-INSIGHT is a Project That Looks at Health Data in Germany to Find Out How Many Patients Suffer From Eye Disease. The Project Also Explores New Ways to Collect and Use Publicly Available Healthcare Information.
Status: Not yet recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 23110
Record Dates: First submitted 2025-12-17; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Neovascular Age-related Macular Degeneration (nAMD); Diabetic Macular Edema (DME); Retinal Vein Occlusion (RVO)
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- nAMD cohort: participants diagnosed with nAMD
  Interventions: Drug: anti-VEGF medication
- DME cohort: participants diagnosed with DME
  Interventions: Drug: anti-VEGF medication
- RVO cohort: participants diagnosed with RVO
  Interventions: Drug: anti-VEGF medication

INTERVENTIONS:
Drug: anti-VEGF medication — according to local label and treating physician

SUMMARY:
The main goal of this study is to find out how common certain eye diseases are in Germany and how they have changed over time. The diseases being studied are:

nAMD (neovascular age-related macular degeneration): a condition that affects the central part of the retina and can cause vision loss in older adults.

DME (diabetic macular edema): a swelling in the central part of the retina caused by diabetes, which can also lead to vision problems.

RVO (retinal vein occlusion): a blockage of the veins in the retina, which can cause sudden vision loss.

Researchers will look at data collected from 2009 to 2024 to see how often these diseases occur (incidence) and how many people have them at a given time (prevalence). They will use two large sets of health data from Germany, called FDZ and FDGP.

The main question is: How do the numbers of new and existing cases of nAMD, DME, and RVO compare between the two data sources (FDZ and FDGP) in Germany from 2009 to 2024? The study also wants to find out if factors like age, other health problems, and medications affect how common these eye diseases are.

Another goal is to see how many people with these eye diseases are treated with a type of medicine called anti-VEGF, which is used to slow down or stop vision loss.

In summary, this study will help us understand how these eye diseases affect people in Germany, how they are treated, and whether different groups of people are more likely to get them.

ELIGIBILITY:
Inclusion Criteria:

* At least one diagnosis of nAMD, DME and RVO in the timeframe 01 JAN 2009 until 31 DEC 2024
* nAMD patients aged ≥ 50 years
* DME patients aged ≥18 years
* RVO patients aged ≥18 years
* Participants living in Germany covered by statutory health insurance or private health insurance

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all participants with the diagnosis of nAMD, DME and RVO from the FDZ and FDGP databases between 1 Jan 2009 and 31 Dec 2024
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
incidence of nAMD, DME and RVO of FDZ and FDPG in Germany | 1 Jan 2009 - 31 Dec 2024
  one-year incidence rate is defined as all new patients fulfilling the inclusion and exclusion criteria in each data repository in the respective year for the first time compared to all patients in the repository in the given year.
prevalence of nAMD, DME and RVO in Germany | 1 Jan 2009 - 31 Dec 2024
  one-year prevalence rate is defined as the proportion of patients fulfilling inclusion and exclusion criteria in each data repository in the respective year PLUS patients identified in any previous year in relation to all patients in the repository in the given year.

SECONDARY OUTCOMES:
incidence of nAMD, DME and RVO of FDZ and FDPG in Germany influenced by demographics, comorbidities, medications and data sources | 1 Jan 2009 - 31 Dec 2024
  one-year incidence rate is defined as all new patients fulfilling the inclusion and exclusion criteria in each data repository in the respective year for the first time compared to all patients in the repository in the given year.
prevalence of nAMD, DME and RVO of FDZ and FDPG in Germany influenced by demographics, comorbidities, medications and data sources | 1 Jan 2009 - 31 Dec 2024
  one-year prevalence rate is defined as the proportion of patients fulfilling inclusion and exclusion criteria in each data repository in the respective year PLUS patients identified in any previous year in relation to all patients in the repository in the given year.
Number of patients with nAMD, DME, and RVO treated with anti-VEGF medications | 1 Jan 2009 - 31 Dec 2024
Proportion of patients with nAMD, DME, and RVO treated with anti-VEGF medications | 1 Jan 2009 - 31 Dec 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer Vital GmbH, Leverkusen, Germany

IPD SHARING:
Plan to Share IPD: No
Currently, there is no established plan for the sharing of Individual Patient Data (IPD) from this study. The availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA 'Principles for responsible clinical trial data sharing.' This pertains to the scope, timepoint, and process of data access. As such, Bayer commits to considering requests from qualified researchers for patient- / study-level clinical trial data, and documents from clinical trials involving medicines and indications approved in the US and EU. However, this commitment does not reflect an active IPD sharing plan. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Researchers can use www.vivli.org to request access to IPD and documents from clinical studies to conduct research. Information on Bayer's criteria for listing studies is provided in the member section of the portal.